CLINICAL TRIAL: NCT02715674
Title: Comparison the Effectiveness of Postoperative Incentive Spirometry and Noninvasive Mechanical Ventilation in Patients Following Craniotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, HULYA KAHRAMAN SAH, MD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 41268
Record Dates: First submitted 2016-02-23; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Neoplasms, Intracranial
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group (Placebo Comparator): take 4lt/min oxygen with Plasti-med oxygen therapy mask
  Interventions: Device: Plasti-med oxygen therapy mask
- IS group (Active Comparator): in postoperatively, patients will carry out Plasti-med TRIFLO 5 min per hour for 6 hours.
  Interventions: Device: Plasti-med TRIFLO
- CPAP group (Active Comparator): in postoperatively, patients will carry out 10 cmH2O noninvasive continuous positive airway pressure with BIPAP VISION 5 min per hour for 6 hours.
  Interventions: Device: BIPAP VISION

INTERVENTIONS:
Device: Plasti-med TRIFLO
  Arms: IS group
Device: BIPAP VISION
  Arms: CPAP group
Device: Plasti-med oxygen therapy mask
  Arms: control group

SUMMARY:
This study will compare the effectiveness of postoperative incentive spirometry and noninvasive mechanical ventilation on pulmonary functions after craniotomy in 60 patients. Patients were randomized into a control group (G-K, n:20), an IS group (G-IS, n:20) and a CPAP (continuous positive airway pressure) group (G-CPAP, n:20)

DETAILED DESCRIPTION:
This study will compare the effectiveness of postoperative incentive spirometry and noninvasive mechanical ventilation on pulmonary functions after craniotomy in 60 patients. Patients were randomized into a control group (G-K, n:20), an IS group (G-IS, n:20) and a CPAP (continuous positive airway pressure) group (G-CPAP, n:20).

The investigators included male or female, between 18 and 60 years old, American Society of Anesthesiologists score 1, 2 patients in this study. The investigator excluded patients with significant cardiopulmonary disease like myocardial infarction, obstructive or restrictive pulmonary disease, liver or kidney failure, chest wall deformities, postoperative lack of cooperation from this study. In postoperatively, control group will take 4lt/min oxygen with Plasti-med oxygen therapy mask for 6 hours, IS group will carry out Plasti-med TRIFLO 5 min per hour for 6 hours, CPAP group will carry out 10 cmH2O noninvasive continuous positive airway pressure with BIPAP VISION 5 min per hour for 6 hours. Lung functions and arterial blood gas analysis will be recorded preoperative baseline, postoperative 1st, 6th and 24th hours.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score 1, 2 patients

Exclusion Criteria:

* Patients with significant cardiopulmonary disease like myocardial infarction, obstructive or restrictive pulmonary disease, liver or kidney failure, chest wall deformities, postoperative lack of cooperation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline forced expiratory volume at one second (FEV1) % predicted (no unit) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Spirolab 3 COLOUR LCD device for measurement.

SECONDARY OUTCOMES:
Change from baseline forced vital capacity (FVC) % predicted (no unit) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Spirolab 3 COLOUR LCD device for measurement.
Change from baseline FEV1/FVC ratio (no units) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Spirolab 3 COLOUR LCD device for measurement.
Change from baseline partial arterial oxygen pressure( PaO2) (mmHg) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Cobas B 221 device for measurement.
Change from baseline partial arterial carbondioxide pressure (PaCO2) (mmHg) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Cobas B 221 device for measurement.
Change from baseline power of hydrogen (pH) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Cobas B 221 device for measurement.
Change from baseline arterial oxygen saturation (SaO2) (%) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Cobas B 221 device for measurement.
Change from baseline base excess (BE) (mmol/L) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Cobas B 221 device for measurement.
Change from baseline bicarbonate (HCO3) (mmol/L) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will use Cobas B 221 device for measurement.
Change from baseline PaO2/FiO2 ratio (no units) | preoperative baseline, postoperative 1st, 6th and 24th hours
  The investigators will calculate PaO2/FiO2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem KORKMAZ DILMEN, Asst. Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty Neurosurgery Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No